CLINICAL TRIAL: NCT03686618
Title: A Phase II Study to Establish the Efficacy of Synthetic Human SecretiN in Human Acute Pancreatitis (SNAP) Study
Brief Title: Secretin for Acute Pancreatitis
Acronym: SNAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ChiRhoClin, Inc. (Industry)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01
Record Dates: First submitted 2018-08-24; First posted 2018-09-27 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis | interventions — Secretin

STUDY DESIGN:
Intervention Model Description: The study is not blinded and does not require any randomization codes. Ten patients each will receive one of three treatments for Days 1, 2, and 3:
  1. No secretin - standard of care and observation (Cohort X)
  2. 32 mcg (<50kg) or 40 mcg (≥50kg)IV Bolus every 12 hours (Cohort 1)
  3. 32 mcg (<50kg) or 40 mcg (≥50kg)IV Bolus every 6 hours (Cohort 2)
  4. 32 mcg (<50kg) or 40 mcg (≥50kg)IV Bolus every 4 hours (Cohort 3)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort X (No Intervention): no secretin administered. All observations
- Cohort 1 (Active Comparator): 32 mcg (<50kg) or 40 mcg (≥50kg) secretin two times a day (40 mcg; q 12 hrs)
  Interventions: Drug: Secretin
- Cohort 2 (Active Comparator): 32 mcg (<50kg) or 40 mcg (≥50kg) secretin four times a day (40 mcg; q 6 hrs)
  Interventions: Drug: Secretin
- Cohort 3 (Active Comparator): 32 mcg (<50kg) or 40 mcg (≥50kg) secretin six times a day (40 mcg; q 4 hrs)
  Interventions: Drug: Secretin

INTERVENTIONS:
Drug: Secretin — Drug to stimulate pancreatic secretion
  Other Names: ChiRhoStim®
  Arms: Cohort 1; Cohort 2; Cohort 3

SUMMARY:
Acute pancreatitis is a frequently devastating pancreatic inflammatory process that results in extensive morbidity, mortality, and hospitalization costs. The incidence of acute pancreatitis has been increasing over the last decade with an overall mortality rate of 5%, although it may be as high as 30% in the most severe cases. It was the most common inpatient gastrointestinal diagnosis in 2009, totaling over 270,000 hospitalizations with estimated "inpatient costs" of over 2.5 billion dollars in the United States. However, despite the significant impact to both patients and the healthcare system, there is no proven pharmacologic therapy that improves important clinical outcomes in acute pancreatitis. The release of bicarbonate rich fluid into the pancreatic duct from the ductal cells is an important mechanism to protect against pancreatitis by two distinct mechanisms:

1. "Flushing" activated enzymes out of the pancreas and into the duodenum thereby preventing accumulation of activated enzymes within the pancreatic acinus
2. Directly alkalinizing the acinar cells, which limits intra-acinar cell damage by improving trafficking of inappropriately activated intra-acinar enzymes along the apical membrane.

In addition to standard care, patients will be divided into 4 cohorts. Cohorts 1,2 and 3 will be treated with different doses of intravenous synthetic human secretin. Cohort X will not receive human secretin, but all datapoints and specimens will be collected. The patient cohorts will be entered into the study as follows: Cohort X; Cohort 1; Cohort 2; Cohort 3. 5 patients in each cohort will be evaluated at each center (for a total of n=10 at both centers for each cohort). Dosing will start within 24 hours of hospitalization with no further synthetic human secretin administration beyond Day 3. Patients will continue to be followed for 7 days or until discharge, whichever comes first. Any data recorded to that point would be included in an intent-to-treat analysis. The primary objective is to perform a Phase II Pilot Study to explore the efficacy of intravenous synthetic human secretin as a pharmacologic adjunct to modulate the severity of human acute (non-obstructive) pancreatitis.

DETAILED DESCRIPTION:
This is a prospective, phase II exploratory pilot study using different dose frequencies of intravenous human secretin in patients with non-obstructive, interstitial acute pancreatitis. All enrolled patients will receive standard of care therapy in regard to fluid resuscitation, pain control, CT scan or ultrasound imaging and nutritional support. In addition to standard of care, patients will be divided into 4 cohorts of 10 patients. Cohorts 1,2 and 3 will receive different doses of intravenous synthetic human secretin. Cohort X will not receive drug. Dosing will start within 24 hours of hospitalization with no further secretin administration beyond Day 3. Patients will continue to be followed until discharge. The primary study endpoint will be the decrease in serum C-reactive protein (CRP) level by 50% within 96 hours and/or at discharge compared with CRP level at admission to determine optimal frequency of dosing. Secondary study endpoints will include: 1) Serum measurements of pro- and anti-inflammatory cytokines including sCD40L, EGF, Eotaxin/CCL11, FGF-2, Flt-3 ligand, Fractalkine, G-CSF, GM-CSF, GRO, IFN-α2, IFN-γ, IL-1α, IL-1β, IL-1ra, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p40), IL-12 (p70), IL-13, IL-15, IL-17A, IP-10, MCP-1, MCP-3, MDC (CCL22), MIP-1α, MIP-1β, PDGF-AA, PDGF-AB/BB, RANTES, TGF-α, TNF-α, TNF-β, VEGF, HSP 27, HSP 60, HSP 70, HSP 90 at time of study enrollment, days of secretin administration, 96 hours and at discharge 2) Clinically relevant outcome measures including hemoconcentration (fall in blood urea nitrogen and hematocrit from admission), decrease in patient admission pain scores (visual analogue scale), decrease in systemic inflammatory response, and tolerance of oral nutrition 3) Calculation of the Dynamic Acute Pancreatitis Score - organ failure, systemic inflammatory response syndrome, abdominal pain, requirement for opiates and ability to tolerate oral intake 4) Length of hospitalization, need for intensive care unit transfer, mortality, need for surgical, endoscopic or percutaneous intervention 5) Development of pancreatic necrosis and/or persistent organ failure and 6) Adverse events and 30 day readmission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female ≥18 years of age
2. Patient voluntarily signed written, informed consent agreement.
3. If patient is female and not more than 1 year post-menopausal, or surgically sterile, must use medically accepted form of contraception or abstain from sexual activities during study
4. Patient has acute pancreatitis as defined by the Atlanta Classification of 2012
5. No evidence of obstructive pancreatitis on available cross-sectional imaging

Exclusion Criteria:

1. Pancreatitis with duct obstruction or severe acute pancreatitis defined by Atlanta Classification
2. Pregnant woman, nursing mothers, or women of childbearing potential not on birth control
3. Known adverse reaction to human secretin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in CRP level | 96 hours and through study completion an average of day 7
  Change in serum C-reactive protein (CRP) level by 50% within 96 hours and/or at discharge compared with CRP level at admission to determine optimal frequency of dosing

SECONDARY OUTCOMES:
Pro- and anti-inflammatory markers | Day 1, Day 2, Day 3, 96 hours and through study completion an average of day 7
  Serum measurements of pro- and anti-inflammatory cytokines including sCD40L, EGF, Eotaxin/CCL11, FGF-2, Flt-3 ligand, Fractalkine, G-CSF, GM-CSF, GRO, IFN-α2, IFN-γ, IL-1α, IL-1β, IL-1ra, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p40), IL-12 (p70), IL-13, IL-15, IL-17A,IP-10, MCP-1, MCP-3, MDC (CCL22), MIP-1α, MIP-1β, PDGF-AA, PDGF-AB/BB, RANTES, TGF-α, TNF-α, TNF-β, VEGF, HSP 27, HSP 60, HSP 70, HSP 90 at time of study enrollment, days of secretin administration, 96 hours and at discharge

OTHER OUTCOMES:
Change in Hemoconcentration measurement | 96 hours and through study completion an average of day 7
  Change in hematocrit from admission
Change in Hemoconcentration measurements | 96 hours and through study completion an average of day 7
  Change in blood urea nitrogen from admission
Acute Pancreatitis Activity Score | 96 hours and through study completion an average of day 7
  A cumulative measurement of the following parameters: (as referenced from the CRF) higher values represent worse outcome Organ Failure (number of systems) x 100 (each system) SIRS (number of criteria) x 25 (each criteria) Abdominal Pain (1-10) x 5 Morphine Equivalent Dose (mg) X 5 Tolerating Solid Diet (yes = 0, no = 1) X 40
Overall hospital stay | 96 hours and through study completion an average of day 7
  Length of hospitalization
Rate of Adverse Events | 30 days following the last administration of study treatment
  Will be reported as a rate per cohort.
Readmission Rate | 30 days following the last administration of study treatment
  Rate will be recorded as number of subjects readmitted within 30 days of final study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Gardner, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Institutes of Health. Opportunities and challenges in digestive diseases research: recommendations of the national commission on digestive diseases. March 2009. Retrieved January 29, 2017.
- [Background] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States Part III: Liver, biliary tract, and pancreas. Gastroenterology. 2009 Apr;136(4):1134-44. doi: 10.1053/j.gastro.2009.02.038. Epub 2009 Feb 24. No abstract available. PMID 19245868
- [Background] Forsmark CE, Vege SS, Wilcox CM. Acute Pancreatitis. N Engl J Med. 2016 Nov 17;375(20):1972-1981. doi: 10.1056/NEJMra1505202. No abstract available. PMID 27959604
- [Background] Peery AF, Dellon ES, Lund J, Crockett SD, McGowan CE, Bulsiewicz WJ, Gangarosa LM, Thiny MT, Stizenberg K, Morgan DR, Ringel Y, Kim HP, DiBonaventura MD, Carroll CF, Allen JK, Cook SF, Sandler RS, Kappelman MD, Shaheen NJ. Burden of gastrointestinal disease in the United States: 2012 update. Gastroenterology. 2012 Nov;143(5):1179-1187.e3. doi: 10.1053/j.gastro.2012.08.002. Epub 2012 Aug 8. PMID 22885331
- [Background] Lerch MM, Saluja AK, Runzi M, Dawra R, Saluja M, Steer ML. Pancreatic duct obstruction triggers acute necrotizing pancreatitis in the opossum. Gastroenterology. 1993 Mar;104(3):853-61. doi: 10.1016/0016-5085(93)91022-a. PMID 7680018
- [Background] Rattner DW. Experimental models of acute pancreatitis and their relevance to human disease. Scand J Gastroenterol Suppl. 1996;219:6-9. doi: 10.3109/00365529609104991. PMID 8865463
- [Background] Hegyi P, Pandol S, Venglovecz V, Rakonczay Z Jr. The acinar-ductal tango in the pathogenesis of acute pancreatitis. Gut. 2011 Apr;60(4):544-52. doi: 10.1136/gut.2010.218461. Epub 2010 Sep 28. PMID 20876773
- [Background] Grady T, Saluja A, Kaiser A, Steer M. Edema and intrapancreatic trypsinogen activation precede glutathione depletion during caerulein pancreatitis. Am J Physiol. 1996 Jul;271(1 Pt 1):G20-6. doi: 10.1152/ajpgi.1996.271.1.G20. PMID 8760102
- [Background] Prinz RA. Mechanisms of acute pancreatitis. Vascular etiology. Int J Pancreatol. 1991 Summer;9:31-8. doi: 10.1007/BF02925576. PMID 1744444
- [Background] Hegyi P, Rakonczay Z Jr. The role of pancreatic ducts in the pathogenesis of acute pancreatitis. Pancreatology. 2015 Jul;15(4 Suppl):S13-7. doi: 10.1016/j.pan.2015.03.010. Epub 2015 Apr 7. PMID 25921231
- [Background] Song L, Wormann S, Ai J, Neuhofer P, Lesina M, Diakopoulos KN, Ruess D, Treiber M, Witt H, Bassermann F, Halangk W, Steiner JM, Esposito I, Rosendahl J, Schmid RM, Riemann M, Algul H. BCL3 Reduces the Sterile Inflammatory Response in Pancreatic and Biliary Tissues. Gastroenterology. 2016 Feb;150(2):499-512.e20. doi: 10.1053/j.gastro.2015.10.017. Epub 2015 Oct 23. PMID 26526716
- [Background] Vege SS, Atwal T, Bi Y, Chari ST, Clemens MA, Enders FT. Pentoxifylline Treatment in Severe Acute Pancreatitis: A Pilot, Double-Blind, Placebo-Controlled, Randomized Trial. Gastroenterology. 2015 Aug;149(2):318-20.e3. doi: 10.1053/j.gastro.2015.04.019. Epub 2015 Jun 23. PMID 26112745
- [Background] Noel P, Patel K, Durgampudi C, Trivedi RN, de Oliveira C, Crowell MD, Pannala R, Lee K, Brand R, Chennat J, Slivka A, Papachristou GI, Khalid A, Whitcomb DC, DeLany JP, Cline RA, Acharya C, Jaligama D, Murad FM, Yadav D, Navina S, Singh VP. Peripancreatic fat necrosis worsens acute pancreatitis independent of pancreatic necrosis via unsaturated fatty acids increased in human pancreatic necrosis collections. Gut. 2016 Jan;65(1):100-11. doi: 10.1136/gutjnl-2014-308043. Epub 2014 Dec 10. PMID 25500204
- [Background] Gardner TB, Vege SS, Pearson RK, Chari ST. Fluid resuscitation in acute pancreatitis. Clin Gastroenterol Hepatol. 2008 Oct;6(10):1070-6. doi: 10.1016/j.cgh.2008.05.005. Epub 2008 Jul 10. PMID 18619920
- [Background] Pitchumoni CS, Agarwal N, Jain NK. Systemic complications of acute pancreatitis. Am J Gastroenterol. 1988 Jun;83(6):597-606. PMID 3287900
- [Background] Chey WY, Chang TM. Secretin: historical perspective and current status. Pancreas. 2014 Mar;43(2):162-82. doi: 10.1097/01.mpa.0000437325.29728.d6. PMID 24518494
- [Background] Chey WY, Chang TM. Secretin, 100 years later. J Gastroenterol. 2003;38(11):1025-35. doi: 10.1007/s00535-003-1235-3. PMID 14673718
- [Background] Hegyi P, Rakonczay Z. Insufficiency of electrolyte and fluid secretion by pancreatic ductal cells leads to increased patient risk for pancreatitis. Am J Gastroenterol. 2010 Sep;105(9):2119-20. doi: 10.1038/ajg.2010.191. No abstract available. PMID 20818368
- [Background] Takacs T, Rosztoczy A, Maleth J, Rakonczay Z Jr, Hegyi P. Intraductal acidosis in acute biliary pancreatitis. Pancreatology. 2013 Jul-Aug;13(4):333-5. doi: 10.1016/j.pan.2013.05.011. Epub 2013 Jun 10. PMID 23890129
- [Background] Hegyi P, Petersen OH. The exocrine pancreas: the acinar-ductal tango in physiology and pathophysiology. Rev Physiol Biochem Pharmacol. 2013;165:1-30. doi: 10.1007/112_2013_14. PMID 23881310
- [Background] Ishiguro H, Naruse S, Kitagawa M, Mabuchi T, Kondo T, Hayakawa T, Case RM, Steward MC. Chloride transport in microperfused interlobular ducts isolated from guinea-pig pancreas. J Physiol. 2002 Feb 15;539(Pt 1):175-89. doi: 10.1113/jphysiol.2001.012490. PMID 11850511
- [Background] Ooi CY, Dorfman R, Cipolli M, Gonska T, Castellani C, Keenan K, Freedman SD, Zielenski J, Berthiaume Y, Corey M, Schibli S, Tullis E, Durie PR. Type of CFTR mutation determines risk of pancreatitis in patients with cystic fibrosis. Gastroenterology. 2011 Jan;140(1):153-61. doi: 10.1053/j.gastro.2010.09.046. Epub 2010 Nov 9. PMID 20923678
- [Background] Freedman SD, Kern HF, Scheele GA. Pancreatic acinar cell dysfunction in CFTR(-/-) mice is associated with impairments in luminal pH and endocytosis. Gastroenterology. 2001 Oct;121(4):950-7. doi: 10.1053/gast.2001.27992. PMID 11606508
- [Background] Behrendorff N, Floetenmeyer M, Schwiening C, Thorn P. Protons released during pancreatic acinar cell secretion acidify the lumen and contribute to pancreatitis in mice. Gastroenterology. 2010 Nov;139(5):1711-20, 1720.e1-5. doi: 10.1053/j.gastro.2010.07.051. Epub 2010 Aug 3. PMID 20691184
- [Background] Hegyi P, Maleth J, Venglovecz V, Rakonczay Z Jr. Pancreatic ductal bicarbonate secretion: challenge of the acinar Acid load. Front Physiol. 2011 Jul 14;2:36. doi: 10.3389/fphys.2011.00036. eCollection 2011. PMID 21808623
- [Background] Goldenberg DE, Gordon SR, Gardner TB. Management of acute pancreatitis. Expert Rev Gastroenterol Hepatol. 2014 Aug;8(6):687-94. doi: 10.1586/17474124.2014.907524. Epub 2014 Apr 25. PMID 24766182
- [Background] Morimoto T, Noguchi Y, Sakai T, Shimbo T, Fukui T. Acute pancreatitis and the role of histamine-2 receptor antagonists: a meta-analysis of randomized controlled trials of cimetidine. Eur J Gastroenterol Hepatol. 2002 Jun;14(6):679-86. doi: 10.1097/00042737-200206000-00014. PMID 12072603
- [Background] Uhl W, Buchler MW, Malfertheiner P, Beger HG, Adler G, Gaus W. A randomised, double blind, multicentre trial of octreotide in moderate to severe acute pancreatitis. Gut. 1999 Jul;45(1):97-104. doi: 10.1136/gut.45.1.97. PMID 10369711
- [Background] Andriulli A, Leandro G, Clemente R, Festa V, Caruso N, Annese V, Lezzi G, Lichino E, Bruno F, Perri F. Meta-analysis of somatostatin, octreotide and gabexate mesilate in the therapy of acute pancreatitis. Aliment Pharmacol Ther. 1998 Mar;12(3):237-45. doi: 10.1046/j.1365-2036.1998.00295.x. PMID 9570258
- [Background] Wu BU, Hwang JQ, Gardner TH, Repas K, Delee R, Yu S, Smith B, Banks PA, Conwell DL. Lactated Ringer's solution reduces systemic inflammation compared with saline in patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):710-717.e1. doi: 10.1016/j.cgh.2011.04.026. Epub 2011 May 12. PMID 21645639
- [Background] Levenick JM, Andrews CL, Purich ED, Gordon SR, Gardner TB. A phase II trial of human secretin infusion for refractory type B pain in chronic pancreatitis. Pancreas. 2013 May;42(4):596-600. doi: 10.1097/MPA.0b013e318273f3ec. PMID 23548879
- [Background] Stevens T, Conwell DL, Zuccaro G Jr, Van Lente F, Lopez R, Purich E, Fein S. A prospective crossover study comparing secretin-stimulated endoscopic and Dreiling tube pancreatic function testing in patients evaluated for chronic pancreatitis. Gastrointest Endosc. 2008 Mar;67(3):458-66. doi: 10.1016/j.gie.2007.07.028. PMID 18294508
- [Background] Conwell DL, Zuccaro G Jr, Vargo JJ, Trolli PA, Vanlente F, Obuchowski N, Dumot JA, O'laughlin C. An endoscopic pancreatic function test with synthetic porcine secretin for the evaluation of chronic abdominal pain and suspected chronic pancreatitis. Gastrointest Endosc. 2003 Jan;57(1):37-40. doi: 10.1067/mge.2003.14. PMID 12518128
- [Background] Renner IG, Wisner JR Jr. Ceruletide-induced acute pancreatitis in the dog and its amelioration by exogenous secretin. Int J Pancreatol. 1986 May;1(1):39-49. doi: 10.1007/BF02795238. PMID 3693975
- [Background] Renner IG, Wisner JR Jr, Lavigne BC. Partial restoration of pancreatic function by exogenous secretin in rats with ceruletide-induced acute pancreatitis. Dig Dis Sci. 1986 Mar;31(3):305-13. doi: 10.1007/BF01318123. PMID 2419062
- [Background] Niederau C, Ferrell LD, Grendell JH. Caerulein-induced acute necrotizing pancreatitis in mice: protective effects of proglumide, benzotript, and secretin. Gastroenterology. 1985 May;88(5 Pt 1):1192-204. doi: 10.1016/s0016-5085(85)80079-2. PMID 2984080
- [Background] Evander A, Lundquist I, Ihse I. Influence of gastrointestinal hormones on the course of acute experimental pancreatitis. Hepatogastroenterology. 1982 Aug;29(4):161-6. PMID 6182081
- [Background] Jowell PS, Branch MS, Fein SH, Purich ED, Kilaru R, Robuck G, d'Almada P, Baillie J. Intravenous synthetic secretin reduces the incidence of pancreatitis induced by endoscopic retrograde cholangiopancreatography. Pancreas. 2011 May;40(4):533-9. doi: 10.1097/MPA.0b013e3182152eb6. PMID 21499206
- [Background] Bakker OJ, van Brunschot S, van Santvoort HC, Besselink MG, Bollen TL, Boermeester MA, Dejong CH, van Goor H, Bosscha K, Ahmed Ali U, Bouwense S, van Grevenstein WM, Heisterkamp J, Houdijk AP, Jansen JM, Karsten TM, Manusama ER, Nieuwenhuijs VB, Schaapherder AF, van der Schelling GP, Schwartz MP, Spanier BW, Tan A, Vecht J, Weusten BL, Witteman BJ, Akkermans LM, Bruno MJ, Dijkgraaf MG, van Ramshorst B, Gooszen HG; Dutch Pancreatitis Study Group. Early versus on-demand nasoenteric tube feeding in acute pancreatitis. N Engl J Med. 2014 Nov 20;371(21):1983-93. doi: 10.1056/NEJMoa1404393. PMID 25409371
- [Background] Eatock FC, Chong P, Menezes N, Murray L, McKay CJ, Carter CR, Imrie CW. A randomized study of early nasogastric versus nasojejunal feeding in severe acute pancreatitis. Am J Gastroenterol. 2005 Feb;100(2):432-9. doi: 10.1111/j.1572-0241.2005.40587.x. PMID 15667504

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03686618/Prot_SAP_000.pdf
  • Informed Consent Form: Drug Cohort ICF (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03686618/ICF_001.pdf
  • Informed Consent Form: Observational Cohort ICF (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03686618/ICF_002.pdf